CLINICAL TRIAL: NCT04140656
Title: The Effects of Plantar Sensory Based Physiotherapy Interventions on Balance and Fallings of Nursing Home Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: muyesser cavlak (Other)
Responsible Party: Sponsor-Investigator, muyesser cavlak, Muyesser CAVLAK, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E52392
Record Dates: First submitted 2019-10-04; First posted 2019-10-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Balance; Distorted; Falling
Keywords: elderly; balance; falling; plantar sensitivity; insole

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized controlled clinical trial; by simple randomization method, cases will be divided into two groups. There are 40 elderly people in the nursing home to be studied. Study was planned as group 1 and group 2. 40 minutes / 3 days per week / 8 weeks long program will be applied to both groups. Four weeks after the first measurement, the second measurement was performed. After the second measurement, rehabilitation program was started in both groups. After the 8-week program is finished, the third measurements will be made. After the third measurements, the fourth measurement will be done 4 weeks later for late results. The measurements are as follows: Primary results: electronic pedobarography device for static and dynamic base pressure changes. Biodex balance test for measuring fall risk and static stability.
  For secondary results; 30 second Chair stand test, Berg balance scale, Semmes weinstein monofilament test.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plantar sensitive exercise group (Active Comparator): Plantar sensitive exercises:
  Interventions: Other: Plantar sensitive exercises
- Textured insole group (Active Comparator): Textured insole group
  Interventions: Other: Textured insole

INTERVENTIONS:
Other: Plantar sensitive exercises — Plantar sensitive exercises:
  40 minutes / 3 days per week / 8 weeks Warm up exercise (5 minute) Walking on different 4 different textured floors and hot floor (15 minute) Trying to recognize small objects with the soles of the feet (5min) Seated work with barbed ball and balance pad (5min) Massage to the sole of the foot with different textured fabrics (5min) Cooling exercise (5 min)
  Arms: Plantar sensitive exercise group
Other: Textured insole — Textured insole group.
  Plantar sensitive exercises with insole 40 minutes / 3 days per week / 8 weeks (all exercises will be done with insoles) Warm up exercise (5 minute) Walking on flat ground (15 minute) Exercise with roller under the sole of the foot (5 minute) Seated work with barbed balance pad (5 min) Dorsi flexion and plantar flexion and hip flexion exercises (5min). Cooling exercise (5 min)
  Arms: Textured insole group

SUMMARY:
Aging in all living things is defined as a normal physiological process that causes a decrease in realistic body function. According to the World Health Organization; It is classified as 65 years old and older and 85 years old and older (1). Characteristics of aging; decrease in reserve capacity of organ systems, decrease in homeostatic control, decrease in adaptability to environmental factors, decrease in stress response capacity (3). Stability is defined as postural stimulation against changes in the center of gravity during rest and activity. Postural answers that provide this harmony; vestibular, proprioceptive and visual data in the central nervous system. In older people, static balance can be maintained for a longer period of time, while dynamic balance may deteriorate more quickly. Aging-affected muscle strength, joint mobility, proprioceptive, vestibular and visual loss also make postural control difficult to achieve. Although the physiological mechanism underlying the risk of loss of equilibrium and falls is multifaceted, it is mostly caused by somatosensory sensitivity and decreased neuromuscular capacity (3-5). It has been determined that one third of the elderly individuals living in the society have fallen at least once a year and these rates have been stated to increase to 60% in nursing homes. Falls cause long-term disability, stay in nursing homes, in the absence of a serious injury as a result of falling, there is a fear of falling, which causes a limitation in activities of daily living. Due to the physiology of aging, it is stated that peripheral sensation decreases in older ages (12). Mold showed that bilateral somatosensorial disorder was present in approximately 26% of individuals aged 65-74, 36% of those aged 75-84, and 54% of those aged 85 years (13). In the literature, it was reported that plantar sensory loss in the elderly affects balance, mobility and gait and is a risk factor for falls (14). Different senses can be sensed by sensing receptors during the exercise program to increase sensory perception. Aerobic and strengthening exercise, feedback, virtual reality have been used in the studies on balance and falling seen in the elderly in recent years. However, a program aimed at increasing plantar sensation and it has not been found in the literature. In this study, physiotherapy programs aimed at increasing plantar sensation in the elderly will be compared.

DETAILED DESCRIPTION:
The study is planned to be conducted between the years of 2019-January-2020 for elderly people over 70 years old who live in Küçük Çamlıca Fahrettin Kerim Gökay Nursing Home. The study was planned as a randomized controlled clinical trial; By simple randomization method, cases will be divided into two groups. There are 47 elderly people over 70 years old in the nursing home to be studied. The sample size was planned to be 16 for each group.Group 1 (n:16), group 2 (n:17). 40 minutes / 3 days per week / 8 weeks long program will be applied to both groups. Four weeks after the first measurement, the second measurement was performed. Thus, pilot study was made. After the second measurement, rehabilitation program was started in both groups.After the 8-week program is finished, the third measurements will be made. After the third measurements, the fourth measurement will be done 4 weeks later for late results.The measurements are as follows.

Primary results: electronic pedobarography device for static and dynamic base pressure changes. Biodex balance test for measuring fall risk and static stability. For secondary results; 30 second Chair stand test, Berg balance scale, Semmes weinstein monofilament test.

ELIGIBILITY:
Inclusion Criteria:

* Voluntariness
* 70 years and older
* Cognitive functions are sufficient for communication (MM score 22 and above)
* 20 meters independent walk
* The soles of the soles are at least at the reduced protective sensory level

Exclusion Criteria:

* Severe visual loss
* A history of mental retardation or schizophrenia
* Person has any problems to prevent walking

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Pedobarographic investigation | day 0 (before intervention)
  By means of pressure sensors in force platforms, foot pressure is detected and transferred to computer environment. Static and dynamic measurement is also possible. Plantar pressure can be measured as total and divided areas and it will be combined to report g/cm2. Plantar contact area can be measured as total and divided areas and it will be combined to report cm2.
Pedobarographic investigation | 4 weeks
  By means of pressure sensors in force platforms, foot pressure is detected and transferred to computer environment. Static and dynamic measurement is also possible. Plantar pressure can be measured as total and divided areas and it will be combined to report g/cm2. Plantar contact area can be measured as total and divided areas and it will be combined to report cm2.
Pedobarographic investigation | 12 weeks
  By means of pressure sensors in force platforms, foot pressure is detected and transferred to computer environment. Static and dynamic measurement is also possible. Plantar pressure can be measured as total and divided areas and it will be combined to report g/cm2. Plantar contact area can be measured as total and divided areas and it will be combined to report cm2.
Pedobarographic investigation | 16 weeks
  By means of pressure sensors in force platforms, foot pressure is detected and transferred to computer environment. Static and dynamic measurement is also possible. Plantar pressure can be measured as total and divided areas and it will be combined to report g/cm2. Plantar contact area can be measured as total and divided areas and it will be combined to report cm2.
Biodex Balance System | day 0 (before intervention)
  It is a multi-axis device which objectively measures the balance of the person in static state or under dynamic stress and records the measurement results. The Biodex Balance System permits a 20 ° inclination of the foot platform in all directions. Thus, it provides maximum stimulation of the mechanical sensors in the ankle. Biodex Balance System measurements are calculated in degrees for each direction It can be done by creating a dynamic environment for the measurement of fall risk on the same platform .
Biodex Balance System | 4 weeks
  It is a multi-axis device which objectively measures the balance of the person in static state or under dynamic stress and records the measurement results. The Biodex Balance System permits a 20 ° inclination of the foot platform in all directions. Thus, it provides maximum stimulation of the mechanical sensors in the ankle. Biodex Balance System measurements are calculated in degrees for each direction It can be done by creating a dynamic environment for the measurement of fall risk on the same platform .
Biodex Balance System | 12 weeks
  It is a multi-axis device which objectively measures the balance of the person in static state or under dynamic stress and records the measurement results. The Biodex Balance System permits a 20 ° inclination of the foot platform in all directions. Thus, it provides maximum stimulation of the mechanical sensors in the ankle. Biodex Balance System measurements are calculated in degrees for each direction It can be done by creating a dynamic environment for the measurement of fall risk on the same platform .
Biodex Balance System | 16 weeks
  It is a multi-axis device which objectively measures the balance of the person in static state or under dynamic stress and records the measurement results. The Biodex Balance System permits a 20 ° inclination of the foot platform in all directions. Thus, it provides maximum stimulation of the mechanical sensors in the ankle. Biodex Balance System measurements are calculated in degrees for each direction It can be done by creating a dynamic environment for the measurement of fall risk on the same platform .

SECONDARY OUTCOMES:
Berg Balance Scala | day 0 (before intervention)
  It is a 14-item clinical scale evaluating static and dynamic equilibrium abilities, each section rated from 0 (poor) to 4 (best). The highest score is 56. A score of less than 45 is an indicator of addiction in daily life. Evaluates the level of dependence and / or independence during positions such as standing up from sitting, standing with feet adjacent, standing in tandem position, staying in balance on one leg and ability to change position. The highest scores indicate the best balance score.
Berg Balance Scala | 4 weeks
  It is a 14-item clinical scale evaluating static and dynamic equilibrium abilities, each section rated from 0 (poor) to 4 (best). The highest score is 56. A score of less than 45 is an indicator of addiction in daily life. Evaluates the level of dependence and / or independence during positions such as standing up from sitting, standing with feet adjacent, standing in tandem position, staying in balance on one leg and ability to change position. The highest scores indicate the best balance score
Berg Balance Scala | 12 weeks
  It is a 14-item clinical scale evaluating static and dynamic equilibrium abilities, each section rated from 0 (poor) to 4 (best). The highest score is 56. A score of less than 45 is an indicator of addiction in daily life. Evaluates the level of dependence and / or independence during positions such as standing up from sitting, standing with feet adjacent, standing in tandem position, staying in balance on one leg and ability to change position. The highest scores indicate the best balance score
Berg Balance | 16 weeks
  It is a 14-item clinical scale evaluating static and dynamic equilibrium abilities, each section rated from 0 (poor) to 4 (best). The highest score is 56. A score of less than 45 is an indicator of addiction in daily life. Evaluates the level of dependence and / or independence during positions such as standing up from sitting, standing with feet adjacent, standing in tandem position, staying in balance on one leg and ability to change position. The highest scores indicate the best balance score
30 Second Chair Stand Test | day 0 (before intervention)
  A test that assesses the person's sit-up activity, lower extremity strength and dynamic balance. Number of sitting and getting up in 30 seconds is noted.
30 Second Chair Stand Test | 4 weeks
  A test that assesses the person's sit-up activity, lower extremity strength and dynamic balance. Number of sitting and getting up in 30 seconds is noted.
30 Second Chair Stand Test | 12 weeks
  A test that assesses the person's sit-up activity, lower extremity strength and dynamic balance. Number of sitting and getting up in 30 seconds is noted.
30 Second Chair Stand Test | 16 weeks
  A test that assesses the person's sit-up activity, lower extremity strength and dynamic balance. Number of sitting and getting up in 30 seconds is noted.
Semmes Weinstein Monofilament Test | day 0 (before intervention)
  Consists of 6 different diameter and equal length monofilments. The test of the sense of touch by questioning whether the person feels the monofilament touches while their eyes are closed.
Semmes Weinstein Monofilament Test | 4 weeks
  Consists of 6 different diameter and equal length monofilments. The test of the sense of touch by questioning whether the person feels the monofilament touches while their eyes are closed.
Semmes Weinstein Monofilament Test | 12 weeks
  Consists of 6 different diameter and equal length monofilments. The test of the sense of touch by questioning whether the person feels the monofilament touches while their eyes are closed.
Semmes Weinstein Monofilament Test | 16 weeks
  Consists of 6 different diameter and equal length monofilments. The test of the sense of touch by questioning whether the person feels the monofilament touches while their eyes are closed.

CONTACTS AND LOCATIONS:
Overall Officials: Candan ALGUN, Prof, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)